CLINICAL TRIAL: NCT03140020
Title: Cognition and Functional Connectivity After Elective Treatment of Brain Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Vienna (Other)
Collaborators: Johannes Kepler University of Linz (Other)
Responsible Party: Principal Investigator, Johannes Kepler University Linz, Univ.Prof.Dr. Andreas Gruber, Johannes Kepler University of Linz
Other Study IDs: KLI 597 B27
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Aneurysm
Keywords: aneurysm; cognition; functional connectivity; frontal lobe function; neuropsychological testing; coiling; clipping
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clipping: Clipping of an aneurysm of the anterior communicating artery - A titan clip will be placed round the aneurysm neck to exclude the aneurysm from the bloodflow and prevent fatal subarachnoidal hemorrhage. Patients will undergo baseline structural MRI, task fMRI, rsfMRI, and baseline neuropsychological examinations prior as well as 2 months after microsurgical aneurysm treatment. Furthermore the patients will undergo additional neuropsychological examinations 12 months after long-term recovery from microsurgical treatment.
  Interventions: Procedure: Clipping
- Coiling: Coiling of an aneurysm of the anterior communicating artery - Using a catheter technique the aneurysm dome will be filled up with coils to prevent subarachnoidal hemorrhage. Patients will undergo baseline structural MRI, task fMRI, rsfMRI, and baseline neuropsychological examinations prior as well as 2 months after endovascular aneurysm treatment. Furthermore the patients will undergo additional neuropsychological examinations 12 months after long-term recovery from endovascular treatment.
  Interventions: Procedure: Coiling
- Healthy Controls: Healthy controls will undergo baseline structural MRI, task fMRI, rsfMRI, and baseline neuropsychological examinations prior as well as 2 months after baseline examinations. Furthermore all subjects will undergo additional neuropsychological examinations 12 months after baseline examination.

INTERVENTIONS:
Procedure: Clipping — During the microsurgical operation a titan clip will be placed round the aneurysm neck to exclude the aneurysm from the bloodflow and prevent fatal subarachnoidal hemorrhage.
  Other Names: microsurgical aneurysm clipping
  Groups: Clipping
Procedure: Coiling — Using a catheter technique the aneurysm dome will be filled up with coils to prevent subarachnoidal hemorrhage.
  Other Names: endovascular treatment of brain aneurysms
  Groups: Coiling

SUMMARY:
The aim of this proposal is to investigate the effects of uneventful microsurgical and endovascular treatment of unruptured saccular non-giant anterior communicating artery [ACoA] aneurysms on resting state functional connectivity levels of higher order cognitive networks and to correlate the connectivity levels of these networks with neuropsychological performance and functional outcome.

This study compares two treatment groups and one control group.

DETAILED DESCRIPTION:
The aim of this proposal is to investigate the effects of uneventful microsurgical and endovascular treatment of unruptured saccular non-giant anterior communicating artery [ACoA] aneurysms on resting state functional connectivity levels of higher order cognitive networks and to correlate the connectivity levels of these networks with neuropsychological performance and functional outcome. The investigators' hypothesis is that the functional connectivity of various cognition networks, i.e. cognitive control network, emotion control of cognitive networks, and working memory networks, as assessed by resting state functional magnetic resonance imaging [rsfMRI], can be impaired after uneventful microsurgical and endovascular treatment of unruptured ACoA aneurysms and can be correlated with neuropsychological performance. The investigators propose to investigate 38 patients harboring unruptured ACoA aneurysms and 19 healthy controls over a 36 (until 48) months period. Patients and healthy controls will undergo baseline structural MRI, task fMRI, rsfMRI, and baseline neuropsychological examinations prior as well as 2 months after either microsurgical or endovascular aneurysm treatment or baseline examinations, respectively. Furthermore all subjects will undergo additional neuropsychological examinations 12 months after baseline examination or long-term recovery from microsurgical and endovascular treatment, respectively. The research question is of substantial importance for this patient population, since it is currently incompletely understood how the minor structural brain tissue damages seen after both treatment methods of unruptured ACoA aneurysms translate into the observed neuropsychological deficits - which are often subtle and transient in nature but still insufficiently explained on grounds of morphology and structural connectivity alone. The sensitivity of rsfMRI to depict the functional communication of spatially remote brain regions presents a novel opportunity to investigate these deficits on a whole brain scale by mapping resting state functional connectivity in higher order cognition networks that are thought to be endangered by events related to both microsurgery and embolization. Correlating these data seems promising for several reasons. First, functional connectivity analysis could be correlated with the neuropsychological impairment in various neuropsychiatric disorders and in ischemic stroke. Ischemic damage to the territories supplied by ACoA perforating arteries is involved in many cases of postoperative neuropsychological impairment after ACoA aneurysm treatment. Second, neuropsychological evaluations have become increasingly incorporated into the standard of care in the postoperative follow-up of cerebral aneurysm patients. RsfMRI could serve as a novel adjunct to neuropsychological outcome assessment. Third, the results could add relevant information to the general perception of the role of frontal lobe and forebrain damage in the pathophysiology of neurocognitive impairment. This could have an impact on neurorehabilitation programs to improve neurocognitive outcome and quality of life in this patient population. Forth, the correlation of validated neuropsychological tests with the functional connectivity rsfMRI data would further enhance the role of rsfMRI in neuroscience and its clinical use.

ELIGIBILITY:
Intervention Groups:

Inclusion criteria

* Male or female patients aged > 18 years
* Microsurgical or endovascular treatment of unruptured, saccular, non giant ACoA aneurysm
* Right-handedness
* Compliance (the patients have to be able to lay motionless in a 3 Tesla MR scanner and to cooperate with the examiner during the examination)
* Willingness and competence to sign informed consent form
* German native speaker

Exclusion criteria

* Ruptured ACoA aneurysm
* Previous history of intracranial hemorrhage or serious head injury
* Non-saccular aneurysm [i.e. dissecting, fusiform, mycotic, traumatic]
* Psychiatric or neuropsychological impairment prior to aneurysm treatment
* Current use of any psychotropic drugs except aneurysm treatment related medication
* Severe visual or auditory impairment
* Current pregnancy or breast feeding
* Metallic implants [other than aneurysm clips or coils detailed in the Ethics section] or other contraindications to MRI

Healthy controls:

Inclusion criteria

* Male or female subjects aged > 18 years
* Right-handedness
* Compliance [the patients have to be able to lay motionless in a 3 Tesla MR scanner and to cooperate with the examiner during the examination]
* Willingness and competence to sign informed consent form
* German native speaker

Exclusion criteria

* Major concurrent or previous medical or neurological illness
* Major concurrent or previous psychiatric Axis I disorder according to DSM-5
* Clinically significant abnormal values in laboratory screening or general physical examination
* Current use of any psychotropic drugs
* Previous history of intracranial hemorrhage, serious head injury
* Previous or current substance abuse [except nicotine and caffeine]
* Severe visual or auditory impairment
* Current pregnancy or breast-feeding
* Metallic implants or other contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated in university hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Prefrontal neuronal functional integration measured with fMRI | Changes pre- vs. posttreatment after 2 months

SECONDARY OUTCOMES:
Prefrontal executive functioning measured with neuropsychological tests | Changes pre- vs. posttreatment after 2 months (short-term outcome) and after 12 months (long-term outcome).
Correlation of changes on neuropsychological (executive functioning) and neuronal level (fMRI). | Changes pre- vs. posttreatment after 2 months measured with fMRI correlated with changes in neuropsychological tests after 2 months (short-term outcome) and after 12 months (long-term outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Gruber, MD, Principal Investigator — Johannes Kepler University of Linz
Locations (2):
- Austria (2):
  - Johannes Kepler University Linz, Dept. of Neurosurgery, Linz, Upper Austria
  - Medical University Vienna, Dep. of Neurosurgery, Vienna

IPD SHARING:
Plan to Share IPD: No